CLINICAL TRIAL: NCT04700982
Title: Does the Length of Hospital Stay for Rehabilitation Affect Functional Outcomes in Stroke Patients: A Retrospective Study
Brief Title: Does the Length of Hospital Stay for Rehabilitation Affect Functional Outcomes in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Betül Çiftçi Tepeli, Department of Physiotherapy and Rehabilitation of Kırklareli University, Kırklareli University
Other Study IDs: 94603339-604.01.02
Record Dates: First submitted 2020-12-28; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Stroke
Keywords: Neurological Rehabilitation; Stroke; Rehabilitation Outcome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Based on the length of hospital stay: Based on the length of hospital stay, patients were divided into two groups: hospital stays ≤ 3 months (Group 1) and > 3 months (Group 2).
  Interventions: Other: Based on the length of hospital stay

INTERVENTIONS:
Other: Based on the length of hospital stay — Based on the length of hospital stay, patients were divided into two groups: hospital stays ≤ 3 months (Group 1) and > 3 months (Group 2).Clinical features and functional output will be then compared between the groups.

SUMMARY:
The purpose of this study was to evaluate whether the length of hospital stay for rehabilitation affects functional outcomes of stroke patients.

DETAILED DESCRIPTION:
The medical records of patients who were admitted to a rehabilitation unit were analyzed retrospectively. The functional output, the level of spasticity, and the level of motor development at admission and discharge will be determined using the Functional Independence Measure instrument, the Modified Ashworth Scale, and the Brunnstrom test, respectively. Based on the length of hospital stay, patients will be divided into two groups: hospital stays ≤ 3 months (Group 1) and > 3 months (Group 2). Clinical features and functional output will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* must be able to receive rehabilitation in an inpatient clinic between 2010 and 2013

Exclusion Criteria:

* previous history of stroke,
* other neurological diseases,
* amputation,
* severe arthritis
* undergoing hemodialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a stroke who received rehabilitation in an inpatient clinic between 2010 and 2013
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical features and Functional Independence Measure instrument, the Modified Ashworth Scale, and the Brunnstrom test outcomes will be then compared between the groups. | through study completion, an average of 1 month
  Demographic features, clinical features and Functional Independence Measure (FIM) instrument, the Modified Ashworth Scale (MAS), and the Brunnstrom test outcomes will be documented for all patients. The FIM includes 18 items with higher scores indicating greater independence. The motor development of the upper extremity, hand, and lower extremity will be evaluated using the Brunnstrom test with higher stages indicating greater development. The degree of spasticity of the upper and lower extremity muscles will be assessed using the MAS with high stage indicating greater spasticity.
  All patients will be divided into two groups based on length of hospital stay. Clinical features, demographic features and FIM, MAS, and the Brunnstrom test outcomes will be then compared between the groups. All data for normality were tested with Kolmogorov-Smirnov tests. Mann-Whitney U tests will be used for comparison of the differences between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: betül çiftçi tepeli, Principal Investigator — Kırklareli University School of Health Department of Physical Medicine and Rehabilitiation
Locations (1):
- Kırklareli Univesity, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foulkes MA, Wolf PA, Price TR, Mohr JP, Hier DB. The Stroke Data Bank: design, methods, and baseline characteristics. Stroke. 1988 May;19(5):547-54. doi: 10.1161/01.str.19.5.547. PMID 3363586
- [Background] Balaban B, Tok F, Yavuz F, Yasar E, Alaca R. Early rehabilitation outcome in patients with middle cerebral artery stroke. Neurosci Lett. 2011 Jul 12;498(3):204-7. doi: 10.1016/j.neulet.2011.05.009. Epub 2011 May 11. PMID 21600267
- [Background] Hebert D, Lindsay MP, McIntyre A, Kirton A, Rumney PG, Bagg S, Bayley M, Dowlatshahi D, Dukelow S, Garnhum M, Glasser E, Halabi ML, Kang E, MacKay-Lyons M, Martino R, Rochette A, Rowe S, Salbach N, Semenko B, Stack B, Swinton L, Weber V, Mayer M, Verrilli S, DeVeber G, Andersen J, Barlow K, Cassidy C, Dilenge ME, Fehlings D, Hung R, Iruthayarajah J, Lenz L, Majnemer A, Purtzki J, Rafay M, Sonnenberg LK, Townley A, Janzen S, Foley N, Teasell R. Canadian stroke best practice recommendations: Stroke rehabilitation practice guidelines, update 2015. Int J Stroke. 2016 Jun;11(4):459-84. doi: 10.1177/1747493016643553. Epub 2016 Apr 14. PMID 27079654